CLINICAL TRIAL: NCT00988728
Title: A Multicenter, Randomized, Parallel-Group, Double-blind, Fixed-Dose, 28-Day Trial to Assess the Efficacy and Safety of SCH 900435 Compared With Placebo, Using Olanzapine as an Active Control in Subjects With an Acute Exacerbation of Schizophrenia (GUEST - Glycine Uptake Inhibitor Efficacy and Safety Trial, Phase 2, Protocol No. P06079)
Brief Title: Efficacy & Safety of SCH 900435 in Schizophrenia (Study P06079)(WITHDRAWN)
Acronym: GUEST
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P06079
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — N-methyl-N-(6-methoxy-1-phenyl-1,2,3,4-tetrahydronaphthalen-2-ylmethyl)aminomethylcarboxylic acid; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SCH 900435 (Experimental): SCH 900435 (Org 25935): a Glycine Uptake Inhibitor
  Interventions: Drug: SCH 900435 (Org 25935); Drug: Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Olanzapine (Active Comparator)
  Interventions: Drug: Placebo; Drug: Olanzapine

INTERVENTIONS:
Drug: SCH 900435 (Org 25935) — Oral tablets, containing 8 mg of active substance, two tablets (i.e. 16 mg) to be taken twice daily in the morning after breakfast and in the evening after dinner during 4 weeks.
  Because of double-dummy design, subjects will be administered two tablets in the morning, and two tablets plus one capsule in the evening (in total 4 tablets with SCH 900435 plus 1 capsule with placebo per day).
  Arms: SCH 900435
Drug: Placebo — Oral capsules and tablets containing excipients only.
  Because of the double-dummy design, subjects will be administered one capsule in the evening, plus two tablets in the morning after breakfast and two tablets after dinner.
Drug: Olanzapine — Oral capsules containing 15 mg of active substance, one capsule to be taken once daily after dinner for four weeks.
  Because of double-dummy design, subjects will be administered two tablets in the morning, and two tablets plus one capsule in the evening (in total 4 tablets with placebo plus 1 capsule with olanzapine per day).
  Other Names: Zyprexa®
  Arms: Olanzapine

SUMMARY:
The purpose of this study is to assess whether SCH 900435 (Org 25935) 16 mg twice daily is more effective than placebo in the treatment of patients with schizophrenia, using olanzapine 15 mg once daily as active control.

ELIGIBILITY:
Inclusion Criteria:

* Subjects eligible to participate:

  * present a substantial and recent exacerbation of schizophrenia
  * have responded positively to treatment with an antipsychotic other than clozapine in the past
  * are without adequate treatment for their symptoms, or willing and capable to stop concurrent medication, which appears inadequate to treat their condition, prior to participation

Exclusion Criteria:

* Schizoaffective disorder;
* single episode of schizophrenia in partial remission
* concomitant use of antidepressants, mood-stabilizers (including anticonvulsants) or long-acting sedatives
* substance abuse or dependence (excluding nicotine and caffeine)
* uncompensated medical illness (including clinically relevant eye disorder)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-02; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
The change from baseline of the Positive and Negative Symptoms Scale (PANSS) (total score) | 4 weeks (Day 28)

SECONDARY OUTCOMES:
Change from baseline in PANSS positive and negative subscale scores (in this order) as compared to olanzapine | 4 weeks